CLINICAL TRIAL: NCT03455543
Title: A Multi-Center, Double-Blind, Sham-Controlled, Randomized Trial of Dual Field PEMF Therapy [Provant® Therapy System] in Lower Extremity Painful Diabetic Distal Symmetric Peripheral Neuropathy (DSPN) (The RELIEF Trial)
Brief Title: Dual Field PEMF Therapy in Lower Extremity Painful Diabetic Distal Symmetric Peripheral Neuropathy
Acronym: RELIEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regenesis Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RBI.2017.002
Record Dates: First submitted 2018-02-28; First posted 2018-03-06 (Actual); Results first posted 2020-03-09 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Diabetic Neuropathy Peripheral

STUDY DESIGN:
Intervention Model Description: Two parallel groups, active device group versus sham device group. Subjects will be randomized 1:1 at baseline and treat with active PEMF or sham for 4 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Active and sham devices will look identical. Participants and site staff will be blind to the randomization.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active Group (Experimental): Treatment with active Provant Therapy System
  Interventions: Device: Active Provant Therapy System
- Sham Group (Sham Comparator): Treatment with in-active (sham) Provant Therapy System
  Interventions: Device: Inactive (sham) Provant Therapy System

INTERVENTIONS:
Device: Active Provant Therapy System — Treatment with active Provant Therapy System
  Arms: Active Group
Device: Inactive (sham) Provant Therapy System — Treatment with inactive Provant Therapy System
  Arms: Sham Group

SUMMARY:
Part A of this trial is a multi-center, prospective, double-blinded, sham-controlled, randomized clinical trial. Part A will evaluate PEMF treatment compared to sham treatment in patients with painful diabetic distal symmetric peripheral neuropathy (DSPN) when treatment is administered 30 minutes twice daily through a 120-day period (4 months). Part B is a 8-month open-label active treatment extension period designed to collect longer-term data on pain, medication use, quality of life and safety (Part B).Part B of this trial is a an extension period upon completion of Part A.

DETAILED DESCRIPTION:
Eligible subjects will be entered into a 14-day ePRO diary run-in period to collect average baseline pain scores related to their diabetic neuropathy in the lower extremities, diary compliance, and analgesic consumption (maintenance and prn prescribed peripheral neuropathic pain medication pill counts). Subjects will collect electronic patient-reported outcome (ePRO) data each morning around the same time during the run-in period.

Subjects will return to the clinic at Baseline (Day 0) for review of eligibility, diary compliance, average baseline diabetic neuropathic pain score of ≥4 and <9, and review of stable analgesic pain consumption profile during the 14-day run-in period. Qualified subjects based on diary compliance and average pain score will be randomized 1:1 (active: sham) and will be instructed to self-treat twice daily for 120 days. Subjects will record electronic patient-reported outcome (ePRO) data following each morning treatment for 120 days. Subjects consenting to distal thigh and distal leg skin biopsies during the Screening visit will have biopsies collected and sent to the central laboratory for assessment. All subjects will have baseline assessments conducted.

Subjects will receive a telephone call at Day 7 to ensure compliance to treatment and diary completion, provide follow-up information on the biopsy sites (if applicable), complete a blinding assessment as well as be assessed for safety and concomitant medication changes.

At Month 1 subjects will return to the clinic for evaluation of safety, concomitant medication changes, review device usage and ePRO diary completion, and Patient Global Impression (PGI). Treatment satisfaction will also be assessed.

At Month 2 subjects will return to the clinic for evaluation of safety, concomitant medication changes, treatment satisfaction, review of device usage (reports will be supplied to the site) and ePRO diary completion, quality of life outcomes (WPAIQ and NeuroQoL), Patient Global Impression (PGI), and interim visit measurements of SPP.

At Month 3, subjects will return to the clinic for evaluation of safety, concomitant medication changes, review device usage (reports will be supplied to the site) and ePRO diary completion, and Patient Global Impression (PGI). Treatment satisfaction will also be assessed.

At Month 4 (end of Part A / start of Part B), subjects will return to the clinic for evaluation of safety, treatment satisfaction, review of device usage (reports will be supplied to the site), HbA1c, concomitant medication changes, weight, quality of life outcomes (WPAIQ and NeuroQoL), PGI, final measurements of SPP, NCS, QST and be assessed to determine their Toronto Clinical Neuropathy Score. Those subjects who consented and had biopsies collected at the Enrollment visit, will have their end of study biopsies during this visit and samples sent directly to the central laboratory for assessment. Subjects will return the study device and complete a blinding assessment.

Subjects that complete Part A will continue into the open-label extension period (Part B). All subjects will be reconsented if not completed at a prior visit and given an open-label active device. Subjects will record ePRO data for one week prior to the Month 6, 8, 10, and 12 visits following each morning treatment. Subjects will be reminded of the150-day (Month 5) phone call.

At Month 5, subjects will receive a telephone call to ensure compliance to treatment, and to be assessed for safety and concomitant medication changes.

At Month 6, subjects will receive a telephone call to ensure treatment compliance and collection of diary data, and to assess safety and concomitant medication changes.

At Month 7, subjects will receive a telephone call to ensure treatment compliance, and to assess safety and concomitant medication changes.

At Month 8, subjects will return to the clinic for evaluation of safety, measure QST, treatment satisfaction, review of device usage and collection of diary data, concomitant medication changes, quality of life outcomes (NeuroQoL), and PGI.

At Month 9, subjects will receive a telephone call to ensure treatment compliance, and to assess safety and concomitant medication changes.

At Month 10, subjects will receive a telephone call to ensure treatment compliance and collection of diary data, and to assess safety and concomitant medication changes.

At Month 11, subjects will receive a telephone call to ensure treatment compliance, and to assess safety and concomitant medication changes.

At Month 12 (end of open-label treatment extension), subjects will return to the clinic for evaluation of safety, weight, QST, NCS, TCNSS, PGI, treatment satisfaction, review of device usage and collection of diary data, concomitant medication changes, quality of life outcomes (NeuroQoL), and will return the study device. Subjects who consented and had biopsies collected at the 4 Month visit, will have their end of study biopsies performed during this visit.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 diabetes
* Pain attributed to symmetrical lower extremity diabetic peripheral neuropathy for at least 6 months
* DPN pain over the preceding 24 hours is ≥4 and <9 based on the 11-point NPRS (0-10)
* 22 to 80 years of age
* On stable diabetes treatment
* HbA1c less than or equal to 10%
* No recent changes to analgesic prescriptions
* ABI of ≥0.8 to ≤1.3
* Walks independently
* Willing and able to give consent
* If female, must be post-menopausal, surgically sterile, abstinent or practicing an effective method of birth control
* Can access an internet browser or smart phone

To be randomized after the 14-day run-in period, average pain (NPRS) must be ≥ 4 and < 9 over preceding 7 days and subject must be 70% compliant with ePRO assessments (electronic diary)

Exclusion Criteria:

* Active, open ulcer on either extremity
* Significant peripheral vascular disease
* Venous insufficiency
* History of solid organ transplant or severe renal disease
* Diagnosed with a non-diabetic cause of chronic neuropathy
* Previous or current history of primary or tertiary hyperparathyroidism, hypercalcemia, psychiatric disorder, alcohol dependency, Hepatitis B or C, or HIV infection
* Significant cardiovascular disease
* Uncontrolled medical illness
* Requires or anticipates the need for surgery during the study
* Total foot depth of >8 cm
* Has received any investigational drug or device within 30 days
* Has used systemic corticosteroids within 3 months
* History of malignancy within 5 years in treatment area
* A psychiatric disorder of sufficient severity
* Receiving prn narcotic medications
* History of drug or alcohol abuse within 1 year
* Implanted pacemaker, defibrillator, neurostimulator, spinal cord stimulator, bone stimulator, cochlear implant, or other implanted device with an implanted metal lead(s0
* Pregnant or planning to become pregnant
* Previous treatment with Provant Therapy
* Unwilling to follow instructions or comply with study instructions
* Pain from any other source that could confuse DPN pain assessment
* Clinically significant foot deformity
* Skin condition that could alter peripheral sensations
* Previous surgery to the spine or lower extremity with residual symptoms of pain or difficulty with movement.
* Clinically significant arthropathy

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2019-07-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Physician's Research Group, Mesa, Arizona
  - Valley Clinical Research, Northridge, California
  - Northern California Research, Sacramento, California
  - Diabetes Research Center, Tustin, California
  - Mountain View Clinical Research, Denver, Colorado
  - Lake Internal Medicine Associates, Eustis, Florida
  - Clinical Physiology Associates, Fort Myers, Florida
  - Spotlight Research Center, Miami, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - River Birch Research Alliance, LLC, Blue Ridge, Georgia
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Heartland Research Associate, LLC, Wichita, Kansas
  - Healthcare Research Network, Hazelwood, Missouri
  - The Center for Pharmaceutical Research, LLC, Kansas City, Missouri
  - Palm Research Center, Las Vegas, Nevada
  - Great Lakes Medical Resarch, Westfield, New York
  - Wake Family Medicine, PC, Cary, North Carolina
  - Rainier Clinical Research, Renton, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Protocol Sample Size was anticipated at 170 subjects. The original enrollment target of 170 subjects was exceeded to grant study entry to qualified subjects that completed the 14-day run-in period.
Groups:
- Open-label Extension Group (Part B): Subjects receiving open-label active PEMF therapy in Part B after 17 weeks of randomized treatment in Part A.
Period: Part A: Randomized Treatment (17 Weeks)
Arm/Group | Active Group | Sham Group | Open-label Extension Group (Part B)
Started | 92 | 90 | 0
Completed | 81 | 83 | 0
Not Completed | 11 | 7 | 0
Not completed — Adverse Event | 2 | 5 | 0
Not completed — Withdrawal by Subject | 7 | 2 | 0
Not completed — Physician Decision | 2 | 0 | 0
Period: Part B: Open-label Extension (24 Weeks)
Arm/Group | Active Group | Sham Group | Open-label Extension Group (Part B)
Started | 0 | 0 | 152
Completed | 0 | 0 | 115
Not Completed | 0 | 0 | 37
Not completed — Adverse Event | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 20
Not completed — Lack of Efficacy | 0 | 0 | 7
Not completed — Lost to Follow-up | 0 | 0 | 4
Not completed — Out of window for visits | 0 | 0 | 2
Not completed — Device interfered with home speakers | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Group | Sham Group | Total
Number analyzed (Participants) | 92 | 90 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.27 (10.21) | 62.17 (9.33) | 62.22 (9.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 42 | 92
  Male | 42 | 48 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 15 | 27
  Not Hispanic or Latino | 80 | 75 | 155
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 14 | 29
  White | 74 | 73 | 147
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 92 | 90 | 182

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity
Description: Absolute change in pain intensity as measured by the 11-point, numerical pain rating scale (NPRS) (0-10; where 0=no pain, to 10=worst possible pain).
Time Frame: Baseline through 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Group | Sham Group
Number analyzed (Participants) | 92 | 90
units on a scale | -1.47 (1.845) | -1.25 (2.018)

2. Secondary Outcome: Patients With 2 Point or 30% Reduction in Pain at 4 Months
Description: Percentage of patients who have either a 2 point or 30% reduction in (pain) NPRS at 4 Months.
  Absolute change in pain intensity as measured by the 11-point, numerical pain rating scale (NPRS) (0-10; where 0=no pain, to 10=worst possible pain).
Time Frame: Baseline to 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Active Group | Sham Group
Number analyzed (Participants) | 92 | 90
Participants | 28 | 26

3. Secondary Outcome: Patient Global Impression at 4 Months
Description: Patient Global Impression at 4 Months. The question assesses change since the start of the study on a 7-point scale ("Since the start of the study, how has your diabetic neuropathy in your legs changed?"), and to score it as either very much worse, much worse, minimally worse, no change, minimally improved, much improved or very much improved.
Time Frame: Baseline through 4 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Group | Sham Group
Number analyzed (Participants) | 92 | 90
Participants
  Much Worse | 1 | 2
  Minimally Worse | 3 | 11
  No Change | 24 | 28
  Minimally Improved | 37 | 23
  Much Improved | 16 | 20
  Very Much Improved | 3 | 3
  Not reported | 8 | 3

4. Secondary Outcome: Time to 30% or 2-point Reduction in NPRS, Whichever Comes First, Through 4 Months
Description: Absolute change in pain intensity as measured by the 11-point, numerical pain rating scale (NPRS) (0-10; where 0=no pain, to 10=worst possible pain). Number of participants achieving a 30% or 2-point reduction at or prior to weeks 1, 4, 8, 12 and 17 are displayed below.
Time Frame: Through 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Active Group | Sham Group
Number analyzed (Participants) | 92 | 90
Participants
  Week 1 | 4 | 3
  Week 4 | 18 | 18
  Week 8 | 32 | 27
  Week 12 | 43 | 34
  Week 17 | 45 | 40

5. Secondary Outcome: Change in Neuropathy Related Quality of Life (NeuroQoL) Between Baseline and End of Treatment at 4 Months.
Description: A validated set of health-related quality of life measures that are domain specific.Subjects will completed 6 domains: (1) Pain, (2) Lost/Reduced Feeling, (3) Diffuse Sensory Motor Symptoms, (4) Restrictions in Activities of Daily Living, (5) Disruptions in Social Relationships, and (6) Emotional Distress.The short forms were completed by the subject at the Enrollment Visit and end of study visit (Day 121). Each question in the domain was rated on a symptom scale from 1 (never) to 5 (all the time) and a bothersome scale from 1 (none) to 3 (very much).
  The total score for the domain was calculated by multiplying the symptom score by the bothersome score. The scale range is from 1 to 15 where the minimum (best/least symptomatic) score is 1 and the maximum (worst/most symptomatic) score is 15. The mean change from Baseline to month 4 is displayed below.
Time Frame: Baseline to 4 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active Group | Sham Group
Number analyzed (Participants) | 92 | 90
units on a scale
  (1) Pain | -1.66 [-2.22 to -1.11] | -1.52 [-2.13 to -0.91]
  (2) Lost/Reduced Feeling | -1.03 [-1.67 to -0.40] | -1.42 [-2.16 to -0.68]
  (3) Diffuse Sensory Motor Symptoms | -0.92 [-1.53 to -0.30] | -0.79 [-1.48 to -0.09]
  (4) Restrictions in Activities of Daily Living | -1.66 [-2.38 to -0.93] | -2.38 [-3.16 to -1.60]
  (5) Disruptions in Social Relationships | -1.31 [-1.99 to -0.62] | -1.99 [-2.70 to -1.29]
  (6) Emotional Distress | -1.12 [-1.68 to -0.55] | -1.63 [-2.33 to -0.93]

6. Secondary Outcome: Change is Skin Perfusion Pressure (SPP) for Baseline to End of Treatment at 4 Months
Description: SPP was measured at two locations on each foot (dorsal right and left and plantar right and left). Mean change displayed from Baseline to 4-months displayed below.
  SPP measures pressure in mmHg; an increase in pressure is favorable.
  * Normal SPP: 50 mmHg to 100 mmHg
  * Marginal Ischemia SPP: 30 mmHg to 50 mmHg
  * Critical Limb Ischemia / PAD SPP: < 30 mmHg
Time Frame: Baseline to 4 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Active Group | Sham Group
Number analyzed (Participants) | 92 | 90
mmHg
  Dorsal - Left | -0.25 (34.22) | 3.27 (33.82)
  Dorsal - Right | -0.74 (35.18) | 2.93 (25.83)
  Plantar - Left | 6.37 (27.72) | -1.84 (28.87)
  Plantar - Right | 2.12 (21.05) | -2.51 (23.66)

7. Secondary Outcome: Changes in Nerve Conduction Studies of Velocity Between Baseline and End of Treatment at 4 Months.
Description: Using the NC-stat DPNCheck, the sural nerve conduction velocity was recorded on the right and left legs. An increase in velocity would suggest DPN improvement. The mean change from Baseline to 4-months is displayed below.
Time Frame: Baseline to 4 Months
Measure: Mean (Standard Deviation); unit: m/s (velocity)
Arm/Group | Active Group | Sham Group
Number analyzed (Participants) | 92 | 90
m/s (velocity)
  Velocity (uv) - Left | -4.15 (20.45) | -5.12 (22.25)
  Velocity (uv) - Right | -1.11 (18.18) | -5.06 (20.94)

8. Secondary Outcome: Changes in Quantitative Sensory Testing (QST) Between Baseline and End of Treatment at 4 Months.
Description: Contact thermal stimulation will be delivered using the Medoc Ltd. Q-Sense system to assess cool sensation threshold, warm sensation threshold and heat pain threshold modalities using the method of limits. Within the cool and warm sensation modalities, the trial is repeated 4 times on each foot and 3 times on each foot for heat pain threshold modality. The cool thermal testing will be conducted prior to the warm and heat pain thermal testing.
  Mean change from baseline to 4-months displayed below.
Time Frame: Baseline to 4 months
Measure: Mean (Standard Deviation); unit: Temperature in degrees C
Arm/Group | Active Group | Sham Group
Number analyzed (Participants) | 92 | 90
Temperature in degrees C
  Cold - Right | 0.57 (3.32) | -0.21 (3.07)
  Cold - Left | 0.08 (3.25) | 0.02 (2.85)
  Warm - Right | -0.58 (3.70) | -0.54 (4.07)
  Warm - Left | -0.53 (4.25) | 0.01 (4.41)
  Pain - Right | -0.29 (3.21) | -0.75 (3.10)
  Pain - Left | -0.62 (3.23) | -0.23 (2.97)

9. Other Pre Specified Outcome: Exploratory Endpoint: Changes in the Work Productivity and Activity Impairment Questionnaire (WPAIQ) (Questions 2-4)
Description: The Work Productivity and Activity Impairment Questionnaire (WPAIQ) is a validated 6 question assessment tool that measures time missed from work, impairment of work and regular activities due to their health problem. Subjects are asked if they are working (Question 1), and if answer is yes, subjects are asked about the effect their diabetic neuropathy (DN) has on their ability to work and perform regular activities in the past 7 days.
  Mean change from Baseline to 4-months are displayed below (Questions 2-4) for subjects that responded "Yes" to working in Question 1. Questions 2-4 are answered in number of hours.
Time Frame: Baseline to 4 Months
Population: Includes only subjects that indicated they were working at the Enrollment Visit (Question 1).
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Active Group | Sham Group
Number analyzed (Participants) | 29 | 18
Hours
  Work hours missed in past 7 days due to DN | 0.12 (2.96) | 0.33 (1.89)
  Work hours missed in past 7 days not due to DN | 0.60 (9.17) | 2.61 (9.38)
  Hours worked in past 7 days | -0.48 (10.62) | -2.11 (20.80)

10. Other Pre Specified Outcome: Exploratory Endpoint: Changes in Intraepidermal Nerve Fiber Density (IENFD) at the Distal Thigh and Distal Leg - Part A
Description: Optional two 3 mm punch skin biopsies will be performed at baseline and end of treatment to assess IENFD. At the Enrollment Visit, one biopsy will be obtained at the distal leg, 10 cm above the lateral malleolus on the right leg and a second biopsy will be obtained at the distal thigh, 10 cm above the superior margin of the patella on the lateral right leg. At the end of Part A study visit Month 4 (Day 121), a second set of biopsies will be obtained lateral to the baseline biopsies and shipped overnight to the central lab.
  For Active Group and Sham Group displayed below, result are the change in nerve fiber density from Baseline to Month 4.
Time Frame: Baseline to Month 4
Measure: Mean (Standard Deviation); unit: nerve fiber density in fibers/mm
Arm/Group | Active Group | Sham Group
Number analyzed (Participants) | 32 | 38
nerve fiber density in fibers/mm
  Right Distal Leg | -0.12 (1.60) | 0.73 (2.33)
  Right Distal Thigh | 0.64 (2.93) | 1.68 (2.63)

11. Other Pre Specified Outcome: Exploratory Endpoint: Change in Pain Intensity During Part B
Description: Absolute change in pain intensity as measured by the 11-point, numerical pain rating scale (NPRS) (0-10; where 0=no pain, to 10=worst possible pain). Results below display the change from Baseline to Month 12 for subjects that participated in the open-label extension (Part B), stratified by their original randomization in Part A.
Time Frame: Baseline through 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Group | Sham Group
Number analyzed (Participants) | 72 | 80
units on a scale | -2.96 (2.38) | 2.49 (2.38)

12. Other Pre Specified Outcome: Exploratory Endpoint: Changes in Nerve Conduction Studies of Velocity During Part B
Description: Using the NC-stat DPNCheck, the sural nerve conduction velocity was recorded on the right and left legs. An increase in velocity would suggest DPN improvement. Results below display the mean change in velocity and from Baseline to Month 12 for subjects that participated in the open-label extension (Part B), stratified by their original randomization in Part A.
Time Frame: Baseline to Month 12
Measure: Mean (Standard Deviation); unit: m/s (velocity)
Arm/Group | Active Group | Sham Group
Number analyzed (Participants) | 72 | 80
m/s (velocity)
  Velocity (m/s) - Left | -11.9 (26.0) | -8.64 (24.7)
  Velocity (m/s) - Right | -9.48 (19.5) | -6.31 (22.9)

13. Other Pre Specified Outcome: Exploratory Endpoint: Change in Neuropathy Related Quality of Life (NeuroQoL) During Part B
Description: A validated set of health-related quality of life measures that are domain specific.Subjects will completed 6 domains: (1)Pain, (2)Lost/Reduced Feeling, (3)Diffuse Sensory Motor Symptoms, (4)Restrictions in Activities of Daily Living, (5)Disruptions in Social Relationships, and (6)Emotional Distress.The short forms were completed by the subject at the Enrollment Visit, end of study visit (Day 121) and at 12 months. Each question in the domain was rated on a symptom scale from 1 (never) to 5 (all the time) and a bothersome scale from 1 (none) to 3 (very much).
  The total score for the domain was calculated by multiplying the symptom score by the bothersome score. The scale range is from 1 to 15 where the minimum (best/least symptomatic) score is 1 and the maximum (worst/most symptomatic) score is 15.
  Results below display the change from Baseline to Month 12 for subjects that participated in the open-label extension (Part B), stratified by their original randomization in Part
Time Frame: Baseline to Month 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Group | Sham Group
Number analyzed (Participants) | 72 | 80
units on a scale
  (1) Pain | -3.14 (2.33) | -2.88 (3.19)
  (2) Lost/Reduced Feeling | -2.42 (2.99) | -1.96 (4.07)
  (3) Diffuse Sensory Motor | -1.58 (2.78) | -1.04 (3.41)
  (4) Restrictions in Activities | -2.67 (3.61) | -2.14 (4.85)
  (5) Distruptions in Social Relationships | -2.25 (3.73) | -1.73 (3.96)
  (6) Emotional Distress | -1.60 (3.81) | -1.79 (3.58)

14. Secondary Outcome: Changes in Nerve Conduction Studies of Amplitude Between Baseline and End of Treatment at 4 Months.
Description: Using the NC-stat DPNCheck, the sural nerve conduction amplitude was recorded on the right and left legs. An increase in amplitude would suggest DPN improvement. The mean change from Baseline to 4-months is displayed below.
Time Frame: Baseline to 4 Months
Measure: Mean (Standard Deviation); unit: uv (amplitude)
Arm/Group | Active Group | Sham Group
Number analyzed (Participants) | 92 | 90
uv (amplitude)
  Amplitude (m/s) - Left | 1.27 (9.96) | 1.36 (11.63)
  Amplitude (m/s) - Right | 1.95 (10.27) | 1.03 (9.91)

15. Other Pre Specified Outcome: Exploratory Endpoint: Changes in Nerve Conduction Studies of Amplitude During Part B
Description: Using the NC-stat DPNCheck, the sural nerve conduction amplitude was recorded on the right and left legs. An increase in amplitude would suggest DPN improvement. Results below display the mean change in amplitude from Baseline to Month 12 for subjects that participated in the open-label extension (Part B), stratified by their original randomization in Part A.
Time Frame: Baseline to Month 12
Measure: Mean (Standard Deviation); unit: uv (amplitude) and m/s (velocity)
Arm/Group | Active Group | Sham Group
Number analyzed (Participants) | 72 | 80
uv (amplitude) and m/s (velocity)
  Amplitude (uv) - Left | 5.28 (14.4) | 4.42 (14.6)
  Amplitude (uv) - Right | 6.0 (15.3) | 4.28 (14.2)

16. Other Pre Specified Outcome: Exploratory Endpoint: Changes in the Work Productivity and Activity Impairment Questionnaire (WPAIQ) (Questions 5-6)
Description: The Work Productivity and Activity Impairment Questionnaire (WPAIQ) is a validated 6 question assessment tool that measures time missed from work, impairment of work and regular activities due to their health problem. Subjects are asked if they are working (Question 1), and if answer is yes, subjects are asked about the effect their diabetic neuropathy (DN) has on their ability to work and perform regular activities in the past 7 days.
  Mean change from Baseline to 4-months displayed below (Questions 5-6) for subjects that responded "Yes" to working in Question 1. Questions 5 and 6 use a 0-10 scale where 0 = no effect on work and/or daily activities and 10 =DN completely prevented me from working and/or doing daily activities.
Time Frame: Baseline to 4 Months
Population: Includes only subjects that indicated they were working at the Enrollment Visit (Question 1).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Group | Sham Group
Number analyzed (Participants) | 29 | 18
units on a scale
  Effect of DN on work in past 7 days | -0.40 (1.89) | -0.61 (3.01)
  Effect on daily activities in past 7 days | -0.67 (2.19) | -0.59 (2.70)

17. Other Pre Specified Outcome: Exploratory Endpoint: Changes in Intraepidermal Nerve Fiber Density (IENFD) at the Distal Thigh and Distal Leg - Part B
Description: Optional two 3 mm punch skin biopsies will be performed at baseline and end of treatment to assess IENFD. At the Enrollment Visit, one biopsy will be obtained at the distal leg, 10 cm above the lateral malleolus on the right leg and a second biopsy will be obtained at the distal thigh, 10 cm above the superior margin of the patella on the lateral right leg. At the end of Part A study visit Month 4 (Day 121), a second set of biopsies will be obtained lateral to the baseline biopsies and shipped overnight to the central lab. At the end of Part B study visit Month 12 (Day 361), a final set of biopsies will be obtained lateral to the Month 4 biopsies.
  Results displayed are the change in nerve fiber density from Baseline to Month 12 for subjects that participated in the open-label extension (Part B), stratified by their original randomization in Part A.
Time Frame: Baseline to Month 12
Measure: Mean (Standard Deviation); unit: nerve fiber density in fibers/mm
Arm/Group | Open-label Extension Group (Part B)
Number analyzed (Participants) | 57
nerve fiber density in fibers/mm
  Right Distal Leg | .22 (2.17)
  Right Distal Thigh | 1.09 (2.94)

ADVERSE EVENTS:
Time Frame: Part A: 4 months (Baseline to Month 4); Part B: 8 months (Month 4 to Month 12)
Groups:
- Active Group (Part A): Treatment with active Provant Therapy System
  Active Provant Therapy System: Treatment with active Provant Therapy System
- Sham Group (Part A): Treatment with in-active (sham) Provant Therapy System
  Inactive (sham) Provant Therapy System: Treatment with inactive Provant Therapy System
- Open-label Extension Group (Part B): Treatment with open-label active Provant Therapy System during Part B (months 4-12)
Arm/Group | Active Group (Part A) | Sham Group (Part A) | Open-label Extension Group (Part B)
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/90 | 57/152
Serious Adverse Events (participants affected / at risk) | 5/92 | 6/90 | 5/152
Other Adverse Events (participants affected / at risk) | 0/92 | 0/90 | 0/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Group (Part A) (N=92) | Sham Group (Part A) (N=90) | Open-label Extension Group (Part B) (N=152)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Pancreatitis
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) — Dehydration
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Congestive heart failure
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) — peripheral vascular disease NOS
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) — COPD exacerbation
Subdural heamatoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Hematoma subdural
seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Seizures
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Sepsis
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) — adenocarcinoma gastric
pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — pneumonia
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Infusion related reaction
abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — right upper quadrant pain
rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — rib fracture
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) — Goitre
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Diverticulum
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Small intestinal obstruction
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) — Chest pain
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Malignant melanoma in situ
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Ischaemic stroke

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication Rights. Independent analysis and/or publication of data generated or arising from the performance of this Agreement is not permitted without the prior written consent of Regenesis. Such consent may be contingent on Regenesis' review and approval of any proposed analysis and manuscript. Institution will retain the right to review and analyze the database created from this study for its own scientific purposes so long as such scientific purposes are non-commercial in nature.

DOCUMENTS (2):
  • Study Protocol (2018-07-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT03455543/Prot_001.pdf
  • Statistical Analysis Plan (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT03455543/SAP_002.pdf